CLINICAL TRIAL: NCT02264847
Title: Trigger or Not to Trigger? : An Answer for an Old Question
Brief Title: Human Chorionic Gonadotrophin & Trigger
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assistant Professor of Obstetrics & Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5102014; A5102014 (Other: Cairo University)
Record Dates: First submitted 2014-10-04; First posted 2014-10-15 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Ovulation Disorder
Keywords: Clomiphene Citrate; Ovulation trigger; Human chorionic gonadotrophin
MeSH Terms: interventions — Chorionic Gonadotropin; Clomiphene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clomiphene citrate plus hCG (Active Comparator): Women will receive clomiphene citrate from day 2 to day 6 of the cycle with a starting dose of 100 mg daily. If no response could be observed, the daily dose of clomiphene citrate in subsequent cycles will be increased by 50 mg until a response will be obtained or a maximum daily dose 200 mg of clomiphene citrate will be used. Once a follicle will reach more than 18 mm in size . Women will receive 5,000 IU human chorionic gonadotrophin trigger in the morning between 9 and 10 a.m. and the couple will be advised to have intercourse the following night, about 36 hours later.
  Interventions: Drug: Human chorionic gonadotrophin
- Clomiphene Citrate alone (Active Comparator): Women will receive clomiphene citrate from day 2 to day 6 of the cycle with a starting dose of 100 mg daily. If no response will be observed, the daily dose of clomiphene citrate in subsequent cycles will be increased by 50 mg until a response will be obtained or a maximum daily dose 200 mg of clomiphene citrate will be used. Once a follicle will reach more than 18 mm in size , the women will be advised to have intercourse frequently over the next few days.
  Interventions: Drug: clomiphene citrate alone

INTERVENTIONS:
Drug: Human chorionic gonadotrophin — Once a follicle reached more than 18 mm in size,women assigned to group (1) received 5,000 IU hCG trigger in the morning between 9 and 10 a.m. and the couple were advised to have intercourse the following night, about 36 hours later.
  Other Names: hCG
  Arms: Clomiphene citrate plus hCG
Drug: clomiphene citrate alone — clomiphene citrate alone without hCG trigger
  Arms: Clomiphene Citrate alone

SUMMARY:
In women being treated with medicines to help eggs to grow (called ovulation induction), The investigators wish to know whether adding medicines (called ovulation triggers) that help to release the egg (ovulation) would lead to more women having babies without causing harm compared with not giving them ovulation triggers.

DETAILED DESCRIPTION:
Women will be treated with clomiphene citrate to help eggs to develop to additionally receive a medicine (urinary hCG) to trigger their release or to receive no additional treatment. the investigators tried to determine the benefits and harms of administering an ovulation trigger to anovulatory women receiving treatment with ovulation-inducing agents in comparison with spontaneous ovulation following ovulation induction. so we will have comparison between 2 groups, group 1 will receive clomiphene citrate and trigger ovulation by human chorionic gonadotrophin and group 2 will receive clomiphene citrate with no drug to trigger ovulation.

ELIGIBILITY:
Inclusion Criteria:

1. Normoprolactinemic and normogonadotropic (WHO class II ovarian dysfunction )
2. Primary infertility with oligomenorrhea (bleeding intervals between 35 days and 6 months) or amenorrhea (bleeding interval more than 6 months)
3. Age 18-40 years
4. Duration of primary infertility more than2 years
5. No history of ovulation induction treatment
6. No history of thyroid disease
7. Normal results on hysterosalpingogram
8. Husband with normal semen analysis

   -

Exclusion Criteria:

1. Ovarian cyst
2. Endometrioma
3. Liver disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Ovulation rate | 1 year
  Collapse of the leading follicle with irregular shape, Appearance of the corpus luteum with diffuse internal echoes. Presence of fluid in the pouch of Douglas or hyperechoic endometrium were taken as supporting features.
  Serum progesterone levels of more than 10 ng/mL were considered to be evidence of ovulation.

SECONDARY OUTCOMES:
chemical pregnancy | 1 year
  A positive urine pregnancy test done 7 days after missing the period
Clinical pregnancy | 1 year
  demonstration of a fetal heart beat on transvaginal ultrasound between 6 and 7 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khyatat, M.D., Principal Investigator — Cairo University
Locations (1):
- faculty of medicine , Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] George K, Kamath MS, Nair R, Tharyan P. Ovulation triggers in anovulatory women undergoing ovulation induction. Cochrane Database Syst Rev. 2014 Jan 31;2014(1):CD006900. doi: 10.1002/14651858.CD006900.pub3. PMID 24482059